CLINICAL TRIAL: NCT00928382
Title: A Pilot Study to Explore Serum and Imaging Biomarkers in Patients With Spinal Cord Compression
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090113; 09-C-0113
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: Cancer; Spine Metastasis
Keywords: Spinal Cord; Healthy Volunteer; Metastasis; Samples; Spinal Cord Vertebrae; Cancer; HV
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
One of the complications of having cancer in the spinal vertebrae is that it can spread and lead to compression of the spinal cord. Spinal cord compression is a serious event that needs to be treated quickly in order to prevent permanent damage to the spinal cord and nerves.

* Researchers currently do not have the ability to accurately predict whether cancer of the vertebrae will cause spinal cord compression. It is possible that accurate predictions could allow doctors to treat patients even before they develop symptoms of spinal cord compression, thereby preventing some of the long-term consequences.

Objectives:

* To compare patients with cancer of the spinal vertebrae with and without symptoms of spinal cord compression by looking at markers in the blood and changes on novel magnetic resonance imaging (MRI) techniques that might allow researchers to predict who will experience spinal cord compression before they actually begin to have symptoms.

Eligibility:

* One group of healthy volunteers 18 years of age and older.
* One group of patients 18 years of age and older who have cancer that has spread to the vertebrae without symptoms of spinal cord compression.
* One group of patients 18 years of age and older who have cancer that has spread to the vertebrae with symptoms of spinal cord compression.

Design:

* Healthy volunteers:
* Blood will be drawn from each volunteer for initial tests and for more specific biomarker tests.
* Comprehensive MRI of the spine, followed by a special type of MRI called diffusion tensor imaging (DTI). It is believed that DTI may be even more sensitive in revealing spinal cord abnormalities than regular MRI sequences.
* Patients with cancer of the vertebrae:
* Researchers will obtain information such as pathology reports, laboratory results, diagnosis and treatment history, physical exam (PE) information, results of scans such as x-rays, MRI, computerized tomography (CT), and positron emission tomography (PET), and planned treatment details.
* Additional blood samples will be taken for specific biomarker tests.
* Questionnaire about pain, unusual sensations or numbness, bladder or bowel problems, and mobility.
* Comprehensive MRI of the spine, followed by a DTI.
* Patients who appear to have symptoms of spinal cord compression will be offered standard radiation treatment.

DETAILED DESCRIPTION:
Background:

* Metastatic Epidural Spinal Cord Compression (MESCC) is an acute and common complication with grave prognosis.
* Biomarkers for early detection and prediction of outcome in these patients may allow a more objective treatment decision algorithm and hopefully change the unfortunate outcome described.
* Serum S-100b, NSE and GFAP and Plasma NF-H are surrogates for neuronal damage in humans and animal models.
* Diffusion tensor imaging (DTI) has been used in brain disorders, in predicting Spinal Cord Injury outcome in animal models, and was found to be beneficial in detecting spinal cord abnormalities in human subjects with acute and slowly progressive cord compression.

Objectives:

* To compare and evaluate the feasibility and reproducibility of DTI of the spinal cord in healthy participants, to optimize the DTI Images and determine normal spine DTI values,
* To describe normal variations of serum/plasma and imaging biomarkers in healthy participants and compare these with serum/plasma and imaging biomarkers values in patients with vertebral metastases with and without spinal cord compression.
* To detect differences in the serum/plasma and imaging biomarkers in patients with vertebral metastases with and without spinal cord compressions.
* To correlate serum/plasma and imaging biomarkers differences with clinical outcomes of patients with vertebral metastases with spinal cord compression (pain, ambulation, continence and survival at 1, 3, 6 and 12 months from radiotherapy).

Eligibility:

* Healthy volunteers with no prior history or concomitant central nervous system injury or inflammatory disease, prior or planned brain or spinal cord radiation therapy or surgical procedure and with no contraindication for MR scanning.
* Patients with metastatic cancer in the spinal vertebrae, with or without spinal cord compression and with no prior history or concomitant central nervous system injury or inflammatory disease, brain metastases, prior brain or spinal cord radiation therapy or surgical procedure and with no contraindication for MR scanning.

Design:

* Preliminary DTI studies will be conducted for healthy volunteer participants to determine normal spine DTI values, choose and optimize the scanning protocol, and evaluate the presence of artifacts and reproducibility of the DTI Images. Normal values and variability of serum and plasma biomarkers will be also determined.
* Patient participants with known vertebral bone metastases with or without spinal cord compression will undergo a DTI study along with the standard MRI sequences, used to evaluate MESCC patients. Blood samples for biomarkers will be also collected.
* Patients with documented MESCC, will be treated with standard radiotherapy fields, dose and schedule. Steroid treatment will be used as clinically indicated. All study procedures will be conducted prior to any therapy. Follow- up visits are planned at 1, 3, 6, and 12 months after radiotherapy completion with history and physical, DTI and serum/plasma biomarker evaluations.

ELIGIBILITY:
* ELIGIBILITY CRITEREIA FOR HEALTHY PARTICIPANTS

Inclusion Criteria:

-Age greater than or equal to 18 years

Exclusion Criteria:

* Inability to provide informed consent.
* History or concomitant central nervous system injury or inflammatory disease (such as stroke, trauma or multiple sclerosis).
* History of radiation therapy to CNS.
* History of brain or spinal cord surgical procedure.
* Contraindication for MR scanning:

  * cardiac pacemaker
  * metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their skull
  * severe claustrophobia
  * metallic orthopedic or other implants
* Allergy to MRI contrast agent.
* Compromised renal function (serum creatinine greater than 1.5) unless patient is on dialysis.

ELIGIBILITY CRITERIA FOR PATIENT PARTICIPANTS

Inclusion Criteria:

* Age greater than or equal to 18 years
* Histologically confirmed cancer.
* Metastatic lesions in the spinal vertebrae, confirmed by CT/MRI/Bone Scan.
* An ECOG performance status of 0, 1 or 2
* A life expectancy of greater than 3 months
* The patient has been evaluated by a neurosurgeon and is not considered a candidate for surgery
* The patient must have a primary physician who specializes in oncology and is willing to collaborate with the ROB staff in the clinical management of the patient.

Exclusion Criteria:

* Inability to provide informed consent
* Patients with primary or secondary CNS malignancy.
* History of spinal cord compression.
* History or concomitant central nervous system injury or inflammatory disease (such as stroke, trauma or multiple sclerosis).
* History of radiation therapy to CNS.
* History or planned brain or spinal cord surgical procedure. Cancer chemotherapy, immunotherapy, or investigational agents received during the 7 days prior to study procedures (hormonal therapy is allowed).
* Contraindication for MR scanning:

  * cardiac pacemaker
  * metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain.
  * severe claustrophobia
  * metallic orthopedic or other metal implants
* History of allergy to MRI contrast agent.
* Compromised renal function (serum creatinine greater than 1.5) unless patient is on dialysis.
* Inability to return for follow up visits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03-31; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gabriel K, Schiff D. Metastatic spinal cord compression by solid tumors. Semin Neurol. 2004 Dec;24(4):375-83. doi: 10.1055/s-2004-861532. PMID 15637649
- [Background] Brihaye J, Ectors P, Lemort M, Van Houtte P. The management of spinal epidural metastases. Adv Tech Stand Neurosurg. 1988;16:121-76. doi: 10.1007/978-3-7091-6954-4_4. No abstract available. PMID 3064753
- [Background] Marquardt G, Setzer M, Seifert V. Protein S-100b as serum marker for prediction of functional outcome in metastatic spinal cord compression. Acta Neurochir (Wien). 2004 May;146(5):449-52. doi: 10.1007/s00701-004-0242-3. Epub 2004 Mar 22. PMID 15118880